CLINICAL TRIAL: NCT03161249
Title: Psychoeducative Treatment of First Episode Psychosis With Mobile Training (ThinkApp):Study Protocol for a Randomised Controlled Trial
Brief Title: Psychoeducative Treatment of FEP With Mobile Training. ThinkApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International University of La Rioja (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PsicoApp
Record Dates: First submitted 2017-05-02; First posted 2017-05-19 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Psychosis; Psychological; Therapy
Keywords: first psychotic episode; mobile app intervention
MeSH Terms: conditions — Psychotic Disorders | interventions — Psychotherapy, Group; Control Groups; Therapeutics

STUDY DESIGN:
Intervention Model Description: This is an experimental, randomized and longitudinal study of repeated measures with independent groups (Treatment group or experimental group: EG and control group: CG) which includes pre and post treatment and 6 months follow-up. This randomized clinical trial includes blind evaluators.
Who Masked: Investigator
Masking Description: blind evaluators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Mobile psychotherapy (5 modules) plus treatment as usual
  Interventions: Behavioral: Experimental group
- Control group (Other): Control group: Treatment as usual
  The description of this group, the control group, corresponds to the treatment to receive the usual treatment that is received on a regular basis, we will not perform any additional intervention
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Experimental group — The experimental group receiving mobile treatment: treatment as usual plus a psychotherapy intervention by the telephone app (a total of 5 modules of psychotherapy: psychoeducation plus mindfulness plus alerts plus social wall plus problems solving)
  Other Names: Psychotherapy group (5 modules)
  Arms: Experimental group
Other: Control group — Group that does not receive any treatment added to its usual treatment
  Other Names: Control group, or treatment as usual group
  Arms: Control group

SUMMARY:
The aim of the study is to evaluate the effectiveness of an online intervention through a mobile application, specifically designed for adolescents with a First Psychotic Episode (FEP), as a complement to the pharmacological and therapeutic interventions they receive at their referral center (Treatment as usual). To do this, a longitudinal study will be carried out on patients with FEP and between the ages of 14 and 30, who come to the Child and Adolescent Psychiatry Service of the General Universitarian Hospital "Gregorio Marañón", Psychiatry Department of the Ramon y Cajal Hospital in Madrid and Psychiatry Department of San Joan de Déu in Catalonia. Adolescents and young will be randomly assigned to an experimental group, where they will receive standard treatment plus online intervention, or a control group, where they will receive standard treatment.

This online intervention, the continuation of the work of this same team researcher in the "PIENSA program", aims to address little of the more traditional treatments and treatments such as community functioning, quality of life or affective symptoms. In addition, it will increase disease awareness, which will lead to greater adherence to treatment and fewer relapses and rehospitalizations.

DETAILED DESCRIPTION:
Clinical assessment criteria Data on the major clinical and demographic variables are entered in a data collection form. All patients are assessed at baseline and have been or will be assessed at 3 months and at 6 months after inclusion in the study. All the instruments used in the study have demonstrated appropriate psychometric properties, and were used in many studies

Demographic data Data are collected on age, sex, level of education, living arrangements and employment or educational status.

Assessment of psychotic symptoms are assessed using the Positive and Negative Syndrome Scale. The scale for the assessment of positive symptoms and negative symptoms. Trait and state anxiety will be measured using the State-Trait Anxiety Inventory. The mood is evaluated using the Hamilton Rating Scale for Depression. We measure patient insight into their illness using the Scale to Assess Unawareness of Mental Disorders. We use the Strauss and Carpenter Prognostic Scale. We also assess the overall function of patients using a Spanish version of the Global Assessment of Functioning Scale. The level of functioning was measured using the Children's Global Assessment Scale. We measure this variable using the "Morisky" Medication Adherence Scale. We measure patient functional status using the Functioning Assessment Short Test.

The consumption is measured using the ASI (Addition severity index) scale. The quality of life is measured using the World Health Organization Quality of Life WHOQOL-BREF Questionnaire .In addition, we assess quality of life using the EuroQoL questionnaire.

Mobile Application Android/Ios Mobile app with a web support and administration application, along with a cloud based backend database, which will register fine-grain interactions between the users and the app, in order to make possible the generation of relevant granular data and key performance indicators to support a wide range of further analysis.

This application will be designed and developed using Software Engineering-based Agile Methodologies, under SCRUM principles (empiric control of the development process, using continuous feedback processes). The whole mobile app functionality and its user interfaces and interactions will be designed under the premises of maximizing the User experience, as a factor contributing to the adherence of users to the treatment.

On the security side, all of the communications between the mobile app and the supporting backend will be protected by means of a "SSL" digital certificate on the server, providing end to end encrypted communications

Data Management For security, all data introduce in database will have an internal code, and will be checked by another data manager, in order to guarantee the data security.

Intervention programme

Mobile phone App treatment

The psychoeducational app programme is composed of 5 modules:

* Psychoeducative Module (12 sessions)
* Module of recognition of symptomatology and prevention of relapses
* Module Troubleshooting
* Mindfulness Module
* Module of social skills

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient between 14-30 years
* The presence of at least 1 positive psychotic symptom (delusions or hallucinations) and 1 of the following diagnoses from DSM-5 (Apa., 2013): schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, major depressive disorder with psychotic features, brief psychotic disorder, or psychosis not otherwise specified.
* Be at least two months without presenting acute psychotic symptoms (delusions or hallucination).
* Written consent given by the patient, parents and / or legal representative.(n this case they must accept to participate both, minor and tutor, concretely, the minors since from the age of 14 also have to accept to participate. )
* Access to a smartphone

Exclusion Criteria:

* Abuse and dependence on toxicants (use is accepted).
* Presence of organic diseases of the central nervous system, mental retardation or generalized developmental disorders

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in psychotic symptoms | Change from Baseline psychotic symptoms at 3 months
  Assessment of psychotic symptoms are assessed using the Positive and Negative Syndrome Scale

SECONDARY OUTCOMES:
Change from Baseline in affective symptoms | Change from baseline affective symptoms at 3 months
  The mood was evaluated using the Hamilton Rating Scale for Depression
Change from Baseline in anxiety level | Change from baseline anxiety symptoms at 3 months
  Anxiety is measured using the State-Trait Anxiety Inventory
Change From Baseline in functionality | Change from Baseline functionality at 3 months
  The functionality is measure using Children's Global Assessment Scale
Change From Baseline in functionality II | Change from baseline functionality at 3 months
  The functionality is measure using Global Assessment of Functioning Scale
Change From Baseline in functionality III | Change from baseline functionality at 3 months
  The functionality is measure using Strauss Carpenter Rating Scale
Change from baseline in prognosis I | Change from baseline prognosis at 3 months
  Number of relapses, hospitalizations and visits to the ER.
Change from baseline in drug´s use | Change from baseline drug´s use at 3 months
  The consumption is measured using the ASI (ASI-6 scale)

OTHER OUTCOMES:
Change from baseline in adherence | Change from baseline adherence level at 3 months
  The adherence is measured using Morisky Medication Adherence Scale
Change from baseline in quality of life | Change from baseline quality of life at 3 months
  The quality of life is measured using the World Health Organization Quality of Life WHOQOL
Change from baseline in quality of life II | Change from baseline quality of life at 3 months
  The quality of life is measured using EuroQoL scale

CONTACTS AND LOCATIONS:
Overall Officials: Ana Calvo, PI, Principal Investigator — UNIR
Locations (1):
- Ana Belén Calvo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barbeito S, Sanchez-Gutierrez T, Mayoral M, Moreno M, Rios-Aguilar S, Arango C, Calvo A. Mobile App-Based Intervention for Adolescents With First-Episode Psychosis: Study Protocol for a Pilot Randomized Controlled Trial. Front Psychiatry. 2019 Feb 5;10:27. doi: 10.3389/fpsyt.2019.00027. eCollection 2019. PMID 30804818